CLINICAL TRIAL: NCT02008032
Title: Comparison of Stationary Breast Tomosynthesis and 2-D Digital Mammography in Patients With Breast Augmentation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients accrued.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 13-1861
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Mammogram Scheduled
Keywords: Mammography; Breast; Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): Stationary Breast Tomosynthesis
  Interventions: Device: Stationary Breast Tomosynthesis

INTERVENTIONS:
Device: Stationary Breast Tomosynthesis — The patient will have the SDBT study performed in a similar manner as conventional mammography in the mediolateral oblique and cranio-caudal plane. The participant will stand up and the mammography research technologist, ensuring patient comfort, will assist in positioning their breast in the breast tomosynthesis unit with standard compression. Once positioned, the total scan time is approximately 10 seconds. Both the left and right breast will be imaged. The length of time for the positioning and examination of a subject's breast may vary but it is expected that the entire imaging procedure will take about 5-10 min, including positioning time.

SUMMARY:
Purpose:The aim of this research is to compare the 3D s-DBT (stationary digital breast tomosynthesis) and conventional 2-D digital mammography devices with regards to patient comfort and radiologist preference in women with breast implants.

Participants: Women with breast implants undergoing routine 2-D digital mammography.

Procedures (methods): 50 female subjects with breast implants undergoing conventional screening mammography will be recruited to have a single view s-DBT in the mediolateral projection. We will perform a patient preference study and radiologist reader study composed of radiologists who have experience evaluating tomosynthesis images. A short survey will be given to each patient about their preference in modality with respect to comfort. Each reader will review the images and score the ease of interpretation, and their confidence of interpretation.

DETAILED DESCRIPTION:
Patients will be recruited with assistance from a referring physician and through patients undergoing routine mammography in the breast imaging clinic.

All eligible women will be contacted by letter and/or phone call prior to scheduled mammography appointment to identify if they would be interested in participating in the research study. On the day of their conventional mammographic imaging, the study will be explained, and they will be offered the opportunity to participate. Consent will happen in a private room in the mammography clinic.

Once consent has been signed, a urine sample will be collected from women who can still become pregnant in order to complete a pregnancy test. Women who are pregnant are unable to participate in this study.

Women who consent for the study will be escorted by the research coordinator to a dressing room, where the subject will change into a gown. The research coordinator or research technologist will then escort the participant to the dedicated study room for the imaging exam. The patient will have the SDBT study performed in a similar manner as conventional mammography in the mediolateral oblique and cranio-caudal plane. The participant will stand up and the mammography research technologist, ensuring patient comfort, will assist in positioning their breast in the breast tomosynthesis unit with standard compression. Once positioned, the total scan time is approximately 10 seconds. Both the left and right breast will be imaged. The length of time for the positioning and examination of a subject's breast may vary but it is expected that the entire imaging procedure will take about 5-10 min, including positioning time.

The breast tomosynthesis scan will be acquired at a dose that is equal to or less than a diagnostic mammogram dose. Upon completion of the breast tomosynthesis exam, the research assistant will provide a short survey to be completed by the patient (less than 5 minutes). The survey will include questions such as the comfort level of s-DBT compared to the standard mammography.

The research SDBT exam will NOT be interpreted prior to the patient leaving the clinic. However, since there is theoretically a possibility of detecting an additional lesion not seen on conventional mammography, all images will be reviewed within a week by a qualified breast imaging specialist. If there are lesions of concern, these will be discussed with the referring surgeon or the patient's primary physician.

After completion of the patient acquisition, a reader study will be performed with five qualified radiologists.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 18 years old.
* Able to provide informed consent.
* History of breast augmentation mammoplasty (at least 1 year prior)

Exclusion Criteria:

* Male. (It is uncommon for men to present for breast imaging)
* Less than 18 years of age.
* Patient unable to give consent. Institutionalized subject (prisoner or nursing home patient).
* Any woman who is pregnant or has reason to believe she is pregnant or any woman who is lactating
* Patient with a history of breast cancer (they would not be a screening exam)
* Patient with a known breast cancer (they would not be a screening study)
* Patient with a lump or nipple discharge (diagnostic population)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Receiver Operative Curve (ROC) Area Under the Curve (AUC) (percentage) | 18 months
  Receiver Operative Curve (ROC) Area Under the Curve (AUC) analysis of the stationary breast tomosynthesis (SDBT) system for the the characterization of suspicious breast lesions in comparison to x-ray mammography.

SECONDARY OUTCOMES:
Reader preference - arbitrary units | 18 months
  To evaluate radiologists confidence in evaluating specific lesion characteristics in suspicious breast lesions. Readers will be scored from -3 to +3.
Patient preference - arbitrary units | 18 months
  To evaluate patient preference of screening methods. Preference will be scored from -3 to +3.

CONTACTS AND LOCATIONS:
Overall Officials: Yueh Lee, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospital, Chapel Hill, North Carolina, United States